CLINICAL TRIAL: NCT02987348
Title: Evaluation of the Clinical and Economic Outcomes Associated With Exenatide Versus Basal Insulin in People With Type 2 Diabetes
Brief Title: Clinical Outcomes of Exenatide Versus Basal Insulin
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5551R00010
Record Dates: First submitted 2016-11-24; First posted 2016-12-08 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- exenatide once weekly: type 2 diabetes patients who were first prescribed with exenatide once weekly in the index period identified from CPRD database of UK primary care
  Interventions: Drug: exenatide once weekly
- basal insulin_1: type 2 diabetes patients who were first prescribed with basal insulin in the index period and matched with exenatide once weekly group identified from CPRD database of UK primary care
  Interventions: Drug: basal insulin
- exenatide twice daily: type 2 diabetes patients who were first prescribed with exenatide twice daily in the index period identified from CPRD database of UK primary care
  Interventions: Drug: exenatide twice daily
- basal insulin_2: type 2 diabetes patients who were first prescribed with basal insulin in the index period and matched with exenatide twice daily group identified from CPRD database of UK primary care
  Interventions: Drug: basal insulin

INTERVENTIONS:
Drug: exenatide once weekly — patients received exenatide once weekly treatment under their standard care, no intervention was given by the study investigator
  Other Names: long_acting glucagon-like peptide-1 receptor agonist
  Groups: exenatide once weekly
Drug: exenatide twice daily — patients with exenatide twice daily treatment under their standard care, no intervention was given by the study investigator.
  Other Names: short-acting glucagon-like peptide-1 receptor agonist
  Groups: exenatide twice daily
Drug: basal insulin — patients with basal insulin treatment under their standard care, no intervention was given by the study investigator
  Other Names: long-acting insulins
  Groups: basal insulin_1; basal insulin_2

SUMMARY:
This is a retrospective cohort study based on Clinical Practice Research Datalink (CPRD) database analysis to compare therapy effectiveness, and cost between exenatide and basal insulin in patients with type 2 diabetes.

Type 2 diabetes (T2DM) is a chronic condition characterized by elevated blood sugar levels (hyperglycaemia) that can result in an increased risk of a variety of conditions including heart disease, strokes, kidney failure, blindness and amputation. Whilst initially patients may control their blood sugar by lifestyle modification (diet and exercise), ultimately most will require therapeutic intervention with regimens that increase in complexity as T2DM progresses. Exenatide is a relatively recent anti-diabetic drug which is known to lead to weight loss as well as improved blood glucose control. It has also been associated with reduced heart attacks and strokes. In this study CPRD database will be used to compare outcomes for patients prescribed exenatide compared with those prescribed insulin; a more established treatment for T2DM. In particular changes from baseline in blood sugar control and weight will be considered as the primary outcomes. As the choice to treat with exenatide or insulin will be related to patient characteristics which may in themselves be associated with the outcomes of the study we aim to match study patients on some of these key variables and adjust for others in our analysis.

DETAILED DESCRIPTION:
Objectives of the study To compare changes in HbA1c and weight from baseline in patients initiated exenatide based-therapy regimen with those initiated insulin-based therapy regimen among type 2 diabetes patients who were injectable naïve in primary care in UK. Health care utilization will be calculated for each of the treatment cohorts, and compared.

Data source Patients will be selected from the Clinical Practice Research Datalink (CPRD), a longitudinal, anonymized research database derived from nearly 700 primary-care practices in the UK. These practices are considered representative of the UK as a whole. The primary-care dataset (CPRD GOLD) comprises data on demographics, diagnoses, hospital referrals, prescriptions emanating in primary care, and other aspects of patient care. Approximately 60% of practices participate in a linkage scheme, by which their patient records are linked to other data sources, including the Hospital Episode Statistics (HES) dataset which provides data on all inpatient and outpatient contacts occurring within National Health Service hospitals in England, and the Office for National Statistics (ONS) mortality dataset. Diagnostic information in the CPRD primary-care dataset is recorded using the Read code classification a UK primary-care practice standard. HES inpatient data are recorded using the International Classification of Disease codes, 10th revision (ICD-10); ONS mortality data are recorded using the ICD-10 and ICD-9 classifications.

Patient identification and Method

Patients defined by CPRD as being of acceptable research quality will be classified as having type 2 diabetes if they had a Read code indicative of diabetes and at least one of the following selection criteria applies:

1. more than one diagnostic record exclusively for type 2 diabetes,
2. prescriptions for two or more different classes of non-insulin glucose-lowering therapy,
3. a diagnostic code indicative of type 2 diabetes (regardless of conflicting diagnoses of type 1 or nonspecific diabetes) plus a prescription for a non-insulin glucose lowering therapy.

Two groups of cases will be defined as patients receiving exenatide as monotherapy or in combination with one or more other oral glucose-lowering therapies based on therapy codes recorded within CPRD. The groups will be:

1. exenatide once weekly formulation (Bydureon),
2. exenatide twice daily formulation (Byetta). Patients will be excluded if they had received

1. prior injectable diabetes therapy 2. less than 90 days continuous exposure to the exenatide therapy Control patients will be selected from the pool of type 2 diabetes patients who had a prescription for basal insulin as monotherapy or in combination with one or more other oral glucose-lowering therapies. The same exclusion criteria as that applied to cases was applied, that is

1. prior injectable diabetes therapy
2. less than 90 days continuous exposure to basal insulin

Matching will be performed by direct matching and by propensity score matching at a ratio of 1:1 based on the following criteria:

1. age (±5 years)
2. gender,
3. year of index exposure (±1 year),
4. diabetes duration (±2 years),
5. BMI (±3 kg/),
6. HbA1c [±1% (±11 mmol/mol)
7. Concurrent glucose-lowering medication.

Index date is the initiation of the study drugs between January 2009 and December 2014.

Primary care and secondary contacts will be ascertained from the CPRD GOLD and HES databases respectively. Admissions will be described by number, length of stay and cost. Healthcare resource groups (HRGs) will be assigned to each patient spell and processed using HRG 4 grouper software (National Casemix Office, Winchester, UK). The allocated HRG will then linked to the 2014 National Tariff adjusted for nature of the admission (elective admissions versus emergency) and excess length of stay. Primary care costs were derived from the Units costs of Health and Social Care 2014 Baseline characteristics of patients initiated on either Bydureon/Byetta and basal insulin will be presented for all patients and for those included in the direct matched and propensity score matched analyses. Differences between characteristics will be tested using the t-test for continuous variables and Pearson chi-square test for categorical variables.

Outcomes All patients received standard care, no interventions were given by the study investigator.

The primary outcome will be HbA1c and weight change. Baseline measures will be defined as any measurement between -180 days and baseline. Change will be measured from baseline to 6 months and 12 - 24 months (± 90 days) for those patients remaining on their index regimen.

HbA1c change from baseline at 6 months and 12-24 months will be calculated and differences between treatment groups compared. The proportion of patients for whom HbA1c falls below 7.0% will also be compared.

Weight change from baseline at 6 months and 12-24 months will be calculated and differences between treatment groups compared. Differences will considered as both an absolute and relative change from baseline.

Two composite end points will be considered based on the proportion of patients:

1. reaching a target of HbA1c<=7.0%% with weight reduction
2. reaching a target of HbA1c<=7.0%% with weight reduction ≥5% The proportion of patients reaching these endpoints were compared by chi-square test. Analyses will be performed for all patients and those matched directly and matched by propensity score.

Secondary outcomes - Health service utilisation Rates and costs of health service contacts will be calculated and compared between treatment groups using the Mann-Whitney U-test. Follow up will be defined as time from index date to last prescription date + 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients who initiated therapy with exenatide or basal insulin between 2009 and 2014.

Exclusion Criteria:

* prior injectable diabetes therapy
* less than 365 days between the latter of the patient's CPRD registration date/practice up-to-standard date and study index date.
* less than 90 days continuous exposure to Exenatide or basal insulin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a non-interventional study based on secondary data analysis. Patients received treatment under their standard care, no intervention was given by the study investigator.
  Patients will be identified and included in the study if they were defined by CPRD as being of acceptable research quality and classified as having type 2 diabetes who initiated exenatide or basal insulin as monotherapy or in combination with one or more other oral glucose-lowering therapies between January 2009 and December 2014.
  Exenatide once weekly (Bydureon) and exenatide twice daily (Byetta) are both investigated, and compared with matched basal insulin cohort.
  Patients will be excluded if they had received prior injectable diabetes therapy and had less than 90 days continuous exposure to the study drugs.
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in HbA1c (%) | 6, 12 and 24 months
  Changes in HbA1c at 6 months, 12 months and 24 months after initiation of the treatment with exenatide and basal insulin will be calculated and compared.
Changes from baseline in weight (kg) | 6, 12 and 24 months
  Changes in weight at 6 months, 12 months and 24 months after initiation of the treatment with exenatide and basal insulin will be calculated and compared.
Changes from baseline in composite outcomes of HbA1c<=7.0% and weight reduction | 6, 12 and 24 months
  Changes in composite outcome of HbA1c<=7.0% and any weight reduction or HbA1c<=7.0% and weight reduction>=5% at 6 months, 12 months and 24 months after initiation of the treatment with exenatide and basal insulin will be calculated and compared.

SECONDARY OUTCOMES:
Health care utilization | 12 months
  Costs of health service contacts after initiation of therapy with exenatide and basal insulin will be calculated and compared using the Mann-Whitney U-test.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Currie, Ph.D, Principal Investigator — Pharmatelligence, UK
Locations (1):
- Pharmatelligence, Cardiff, United Kingdom

REFERENCES:
- [Background] Holden SE, Morgan CL, Qiao Q, Jenkins-Jones S, Berni ER, Currie CJ. Healthcare resource utilization and related financial costs associated with glucose lowering with either exenatide or basal insulin: A retrospective cohort study. Diabetes Obes Metab. 2017 Aug;19(8):1097-1105. doi: 10.1111/dom.12916. Epub 2017 Mar 31. PMID 28218819
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4435&filename=D5551R00010_Poster_ADA2016.pdf